CLINICAL TRIAL: NCT02272478
Title: A Trial for Older Patients With Acute Myeloid Leukaemia and High Risk Myelodysplastic Syndrome
Brief Title: Trial to Test the Effects of Adding 1 of 2 New Treatment Agents to Commonly Used Chemotherapy Combinations
Acronym: AML18
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardiff University (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Principal Investigator, Prof Nigel Russell, Prof, Cardiff University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AML18
Record Dates: First submitted 2014-06-10; First posted 2014-10-23 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2019-08

CONDITIONS: Acute Myeloid Leukaemia; Myelodysplastic Syndrome
Keywords: AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Gemtuzumab; CPX-351; Decitabine; vosaroxin; Nuclear Receptor Subfamily 4, Group A, Member 2; Ida-FLAG protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm A (Active Comparator): Patients not known adverse karyotype
  Randomise between
  Daunorubicin 60mg/m2 daily by i.v. infusion on days 1, 3 and 5 (3 doses) Cytosine Arabinoside 100mg/m2 12 hourly by i.v. push on days 1 - 10 inclusive (20 doses) Mylotarg (GO) 3mg/m2 on day 1 of DA chemotherapy
  Versus
  CPX-351 100 units/m2 on days 1, 3 and 5
  Interventions: Drug: Arm A Mylotarg plus DA Versus CPX-351
- Arm B (Active Comparator): Patients with known adverse karyotype
  5 cycles of Vosaroxin and Decitabine therapy
  Interventions: Drug: Arm B Vosaroxin and Decitabine
- Arm C (Active Comparator): Prior to Course 2 - Patients receving DA plus GO in course 1 and MRD positive PC1
  Randomise between
  Daunorubicin 50mg/2 daily by i.v. infusion on days 1, 3 and 5 (3 doses) Cytosine Arabinoside 100mg/m2 12 hourly by i.v.push on days 1 - 8 inclusive (16 doses)
  Versus
  Daunorubicin 50mg/m2 daily by i.v. infusion on days 1, 3 and 5 Cytosine Arabinoside 100mg/m2 12 hourly by i.v. push on days 1 - 8 inclusive Cladribine 5mg/m2 daily on days 1 - 5 inclusive
  Versus Patients aged 60-69 Fludarabine 30mg/m2 daily on i.v. on days 2 - 6 inclusive Cytosine Arabinoside 1g/m2 daily over 4 hours Fludarabine on days 2 - 6 inclusive
  Patients aged 70+ Fludarabine 25mg/m2 daily i.v. on days 2 - 5 inclusive Cytosine Arabinoside 1g/m2 daily over 4 hours Fludarabine on days 2 - 5 inclusive Idarubicin 5mg/m2 i.v. daily on days 3, 4 and 5 (3 doses)
  And Randomisation to receive AC220 or not
  Interventions: Drug: Arm D Small molecule or Not; Drug: Arm C DA V FLAG-Ida V DAC
- Arm D (Active Comparator): Prior to Course 2 - Patients that received DA plus GO in course 1 and MRD negative PC1
  Randomisation to receive AC220 or not
  Interventions: Drug: Arm D Small molecule or Not
- Arm E (Active Comparator): Prior to Course 2 for patients receiving CPX in course 1 and MRD positive PC1
  Randomisation between
  CPX-351 100 units/m2 on days 1, and 3 (CPX 200) versus CPX-351 100 units/m2 on days 1, 3 and 5 (CPX 300)
  Interventions: Drug: Arm E CPX-351 (200 V 300)
- Arm F (Active Comparator): Prior to Course 3 - Patients that received DA plus GO in course 1 and MRD negative PC1
  Randomise between Daunorubicin 50 mg/m2 daily by i.v. infusion on days 1 and 3 (2 doses) Cytosine Arabinoside 100 mg/m2 12-hourly by i.v. push on days 1 - 5 inclusive (10 doses)
  versus
  Intermediate dose Cytarabine (IDAC) schedule Cytosine Arabinoside 1g/m2 daily by 4 hour infusion on days 1- 5 inclusive (5 doses)
  Interventions: Drug: Arm F DA V IDAC

INTERVENTIONS:
Drug: Arm A Mylotarg plus DA Versus CPX-351 — Patients not known to have adverse risk cytogenetics will enter a randomisation comparing DA with Mylotarg (GO) delivered at 3mg/m2 on day 1 of chemotherapy, with CPX-351 on days 1, 3 and 5.
  Other Names: Mylotarg (GO); CPX-351
  Arms: Arm A
Drug: Arm B Vosaroxin and Decitabine — If a patient is known to have adverse risk Cytogenetics at diagnosis they will enter a registration to receive up to 5 courses of Vosaroxin and Decitabine.
  Other Names: Vosaroxin; Decitabine
  Arms: Arm B
Drug: Arm D Small molecule or Not — The randomisation to AC220 or not will take place immediately before course 2 of treatment for patients who have received DA induction +/- Mylotarg, irrespective of residual disease status. Patients allocated to receive AC220 will be randomised in a 1:1 fashion to AC220 or no small molecule with a 1:1 randomisation in patients drawing AC220 between short and long therapy.
  Other Names: No AC220
  Arms: Arm C; Arm D
Drug: Arm C DA V FLAG-Ida V DAC — If a patient is not in CR or CRi after course 1 or is MRD +ve/unknown by flow cytometry they will be eligible to be randomised in a 1:1:1 fashion between DA, FLAG-Ida (or mini FLAG-Ida if 70 years or older) and DAC.
  Other Names: DA; FLAG-Ida; DAC
  Arms: Arm C
Drug: Arm E CPX-351 (200 V 300) — If a patient is not in CR or CRi after course 1 or is MRD +ve/unknown by flow cytometry they will be eligible to be randomised in a 1:1 fashion between CPX given on days 1, 3 and 5 (3 doses) and CPX given on days 1 and 3 (2 doses).
  Other Names: CPX-351
  Arms: Arm E
Drug: Arm F DA V IDAC — Following recovery from course 2, patients in the MRD-ve arm will be randomised between a further 5-day cycle of DA or a cycle of intermediate dose cytarabine (IDAC) as the third chemotherapy course.
  Other Names: IDAC; DA
  Arms: Arm F

SUMMARY:
The AML18 Trial will evaluate several relevant therapeutic questions in Acute Myeloid Leukaemia (AML), as defined by the WHO, and High Risk Myelodysplastic Syndrome. The trial is primarily designed for patients over 60 years considered fit for an intensive chemotherapeutic approach, but younger patients who may not be considered suitable for the concurrent NCRI AML Trial for younger patients may also enter. Patients for whom intensive chemotherapy is not thought suitable may enter the concurrent NCRI trial of less intensive therapy (LI1). Approximately 1600 patients will be recruited.

At entry, a randomisation will compare a standard chemotherapy schedule DA (Daunorubicin/Ara-C) combined with 1 dose of Mylotarg (gemtuzumab ozogamicin, or GO) in course 1 against CPX-351. Patients who have known adverse risk cytogenetics (using Grimwade 2010 classification favourable/intermediate/adverse) at diagnosis may enter a Phase 2 evaluation of the combination of Vosaroxin plus Decitabine. Patients who achieve complete remission (CR) and who are MRD negative by flow cytometry after course one of DA will receive one further course of DA, with a randomisation to receive, either a course of DA or intermediate dose Cytarabine (IDAC) as a third course. Patients who are MRD negative by flow cytometry after course one of CPX-351 will receive up to 2 further course of CPX. Patients who fail to achieve a CR after course 1 of DA or who are MRD positive by flow cytometry or for whom MRD information is not available, are eligible to be randomised to compare DA with DA plus Cladribine (DAC) or FLAG-Ida for up to two courses of therapy. Patients who fail to achieve a CR after course 1 of CPX-351 or who are MRD positive by flow cytometry or for whom MRD information is not available are eligible to be randomised between a second course of standard dose CPX versus a repeat of the course 1 schedule. Patients receiving Vosaroxin and Decitabine are excluded from these post course 1 randomisations .

Following the outcome of course 1, patients who received DA chemotherapy on course 1 will be randomised to receive further chemotherapy with the 2nd generation FLT3 inhibitor AC220. Patients randomised to AC220 will be allocated a maximum of 3 courses (short AC220) or 3 courses plus maintenance for 1 year (long AC220). Patients receiving Vosaroxin and Decitabine are excluded from this randomisation.

Patients will be eligible for a non-intensive allogeneic stem cell transplant if a suitable HLA matched donor is available.

DETAILED DESCRIPTION:
AML18 is a trial primarily for older patients with AML and high risk Myelodysplastic Syndrome (MDS). It offers a randomised controlled Phase II/III trial which uses a factorial design for maximum efficiency to evaluate two induction options followed by treatment with small molecule beyond course 1, and dose intensification for patients without evidence of MRD negativity.

There are five randomised comparisons within the trial:

1. At diagnosis:

   For patients not known to have adverse risk cytogenetics DA chemotherapy plus a single dose of 3 mg/m2 of Mylotarg versus CPX-351. Patients with abnormal LFTs can enter the randomisation but receive DA alone or CPX-351.
2. For patients who received DA chemotherapy but are not in CR or who are MRD +ve, or for whom MRD is not assessable.

   DA versus DAC versus FLAG-Ida
3. All patients at second course who have received DA and have not received Vosaroxin and Decitabine induction AC220 versus no AC220 for a maximum of 3 cycles; then with or without maintenance for 1 year for patients allocated AC220
4. For patients who are in CR or CRi and MRD -ve post course1 and have completed 2 courses of DA DA versus intermediate dose Cytarabine (IDAC)
5. For patients who received CPX-351 chemotherapy but are not in CR or who are MRD +ve, or for whom MRD is not assessable CPX-351 100 units/m2 x 3 doses versus CPX-351 100 units/m2 x 2 doses

The trial will also assess:

* Non-intensive allogeneic stem cell transplant for patients with matched sibling or matched unrelated donors.
* The combination of Vosaroxin and Decitabine for those with known adverse risk cytogenetics at diagnosis

ELIGIBILITY:
Inclusion Criteria

Patients are eligible for the AML18 trial if:

* They have one of the forms of acute myeloid leukaemia, except Acute Promyelocytic Leukaemia as defined by the WHO Classification (Appendix A) this can be any type of de novo or secondary AML - or high risk Myelodysplastic Syndrome, defined as greater than 10% marrow blasts (RAEB-2). (NB patients with prior MDS (>10% blasts, RAEB2) have received azacitidine are not eligible for the trial, but patients with <10% who have failed a hypomethylating agent and developed AML may enter the trial).
* Patients should normally be over the age of 60, but patients under this age are eligible if they are not considered eligible for the MRC AML19 trial please contact the trial team for further information.
* Patients entering the Vosaroxin/Decitabine arm must be over the age of 60 and have known adverse risk cytogenetics.
* They have given written informed consent.
* Serum creatinine ≤ 1.5 × ULN (upper limit of normal)
* Sexually mature males must agree to use an adequate and medically accepted method of contraception throughout the study if their sexual partners are women of child bearing potential (WOCBP). Men should be advised to not father a child while receiving trial treatment. Similarly women must agree to adequate contraceptive measures and avoid becoming pregnant while on protocol treatment. In both males and females these measures must be in place for at least 3 months following completion of Decitabine and at least 6 months after the last administration of Cladribine. The time period following treatment with Decitabine where it is safe to become pregnant is unknown. In the event of pregnancy at any point during the trial, the IMPs should be immediately stopped and the Trial Team should be contacted and pregnancy reporting procedures followed.
* ECOG Performance Status of 0-2

Exclusion criteria

Patients are not eligible for the AML18 trial if:

* They have previously received cytotoxic chemotherapy for AML [Hydroxycarbamide, or similar low-dose therapy, to control the white count prior to initiation of intensive therapy, is not an exclusion]
* They are in blast transformation of chronic myeloid leukaemia (CML)
* They have a concurrent active malignancy excluding basal cell carcinoma
* They are pregnant or lactating
* They have Acute Promyelocytic Leukaemia
* Known infection with human immunodeficiency virus (HIV)
* Patients with prior cumulative anthracycline exposure (from prior treatment of a non AML cancer) of greater than 300 mg/m2 daunorubicin (or equivalent).
* History of myocardial infarction (MI), unstable angina, cerebrovascular accident, or transient ischemic attack (CVA/TIA) within 3 months before entry

Specific exclusion criteria for the Mylotarg Arm

* Pre-existing liver impairment with known cirrhosis
* Total bilirubin > 1.5 x the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) > 2.5 x ULN
* Alanine aminotransferase (ALT) > 2.5 x ULN

Specific exclusion criteria for the Vosaroxin/Decitabine Entry

* Total bilirubin > 1.5 x the upper limit of normal (ULN),
* Aspartate aminotransferase (AST) > 2.5 x ULN
* Alanine aminotransferase (ALT) > 2.5 x ULN
* Left ventricular ejection fraction (LVEF) < 40% by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)]

Specific exclusion criteria for CPX-351 treatment

* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or other copper-metabolism disorder

Specific exclusion criteria for Cladribine

• Patient's serum creatinine must be within the local ULN to enter the randomisation. Patients for whom this is not the case can be randomised between the remaining options.

In addition patients are not eligible for the AC220 randomisation if they have:

Cardiovascular System Exclusion Criteria:

Known serious cardiac illness or medical conditions, including but not limited to:

I. Clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, active myocardial ischemia, or indwelling temporary pacemaker II. Ventricular tachycardia or a supraventricular tachycardia that requires treatment with a Class Ia antiarrhythmic drug (e.g., quinidine, procainamide, disopyramide) or Class III antiarrhythmic drug (e.g., sotalol, amiodarone, dofetilide). Use of other antiarrhythmic drugs is permitted.

III. Use of medications that have been linked to the occurrence of torsades de pointes (see Appendix for the list of such medications) IV. Second- or third-degree atrioventricular (AV) block unless treated with a permanent pacemaker V. Complete left bundle branch block (LBBB) VI. History of long QT Syndrome or a family member with this condition VII. Serum potassium, magnesium, and calcium levels not outside the laboratory's reference range VIII. QTc >450 ms (average of triplicate ECG recordings); a consistent method of QTc calculation must be used for each patient's QTc measurements. QTcF (Fridericia's formula) is preferred. Please see the trial website for QTcF calculator.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2014-10-30 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
Complete remission (CR + CRi) achievement and reasons for failure (for induction questions) | 1 month
Duration of remission, relapse rates and deaths in first CR | 1 month
Toxicity, both haematological and non-haematological | 1 month
Supportive care requirements (and other aspects of health economics) | 6 months

SECONDARY OUTCOMES:
The relevance of the presence of a cytogenetic abnormality in the bone marrow of patients in morphological remission | At study end
The relevance of molecular characteristics and response to treatment | 1 month
To store diagnostic tissue for future research in the AML Tissue Bank | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Nigel Russell, Prof, Principal Investigator — Nottingham University
Locations (87):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Herlev and Gentofte Hospital, Copenhagen
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
  - Roskilde Hospital, Roskilde
- United Kingdom (81):
  - Aberdeen Royal Infirmary, Aberdeen
  - Monklands Hospital, Airdrie
  - Ysbyty Gwynedd Hospital, Bangor
  - Royal United Hospital Bath, Bath
  - Belfast City Hospital, Belfast
  - Birmingham Heartland Hospital, Birmingham
  - Queen Elizabeth Hospital, Birmingham
  - Blackpool Victoria Hospital, Blackpool
  - Ysbyty Glan Clwyd, Bodelwyddan
  - Pilgrim Hospital, Boston
  - Royal Bournemouth General Hospital, Bournemouth
  - Bradford Royal Infirmary, Bradford
  - Bristol Haematology & Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - UHW, Cardiff
  - University Hospital of Wales, Cardiff
  - Cheltenham General Hospital, Cheltenham
  - Countess of Chester Hospital, Chester
  - St Richard's Hospital, Chichester
  - University Hospital of Coventry and Warwickshire, Coventry
  - Derby Teaching Hospital, Derby
  - Russell Hall, Dudley
  - Ninewells Hospital, Dundee
  - Western General Hospital, Edinburgh
  - Royal Devon & Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Hairmyres Hospital, Glasgow
  - The New Victoria Hospital, Glasgow
  - Gloucestershire Royal Hospital, Gloucester
  - Royal Free Hospital, Hamstead
  - Raigmore Hospital, Inverness
  - Ipswich Hospital, Ipswich
  - Crosshouse & Ayr Hospital, Irvine
  - Kettering General Hospital, Kettering
  - Victoria Hospital, Kirkcaldy
  - Forth Valley Royal Hospital, Larbert
  - St Jame's University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Lincoln County Hospital, Lincoln
  - Aintree University Hospital, Liverpool
  - The Royal Liverpool University Hospital, Liverpool
  - Guy's Hospital, London
  - St Bartholomew's Hospital, London
  - St George's Hospital, London
  - The Royal Marsden, London
  - University College London Hospital, London
  - Maidstone District General Hospital, Maidstone
  - Manchester Royal Infirmary, Manchester
  - The Christie Hospital, Manchester
  - Arrowe Park Hospital, Metropolitan Borough of Wirral
  - The James Cook University Hospital, Middlesbrough
  - Milton Keynes, Milton Keynes
  - Freeman Hospital, Newcastle
  - Northampton General Hospital, Northampton
  - Norfolk & Norwich University, Norwich
  - Nottingham University Hospital, Nottingham
  - Royal Oldham Hospital, Oldham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Queen Alexandra Hospital, Portsmouth
  - Whiston Hospital & St Helens, Prescot
  - Queen's Hospital, Romford
  - Salford Royal Hospital, Salford
  - Salisbury District Hospital, Salisbury
  - Wexham Park Hospital, Slough
  - Southampton General Hospital, Southampton
  - Stafford Hospital, Stafford
  - University Hospital of Royal Stoke, Stoke-on-Trent
  - Sunderland Royal Hospital, Sunderland
  - St Helier Hospital, Sutton
  - Singleton Hospital, Swansea
  - Torbay District General Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Hillingdon Hospital, Uxbridge
  - Pinderfields Hospital, Wakefield
  - Sandwell Hospital, West Bromwich
  - Wishaw General Hospital, Wishaw
  - New Cross Hospital, Wolverhampton
  - Worcestershire Royal Hospital, Worcester
  - Worthing Hospital, Worthing
  - York Hospital, York